CLINICAL TRIAL: NCT05870904
Title: A Randomized Clinical Trial To Review The Effectiveness Of Dry Needling Versus Trigger Point Compression Release Among Patients With Neck Pain
Brief Title: Dry Needling & Trigger Point Compression Release in Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Health Education Research Foundation (HERF) (Other)
Responsible Party: Principal Investigator, Mamoona Tasleem Afzal, Senior Lecturer, Health Education Research Foundation (HERF)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 070/BPMI/ Saad Tariq DPT
Record Dates: First submitted 2023-04-26; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Neck Pain; Trigger Point Pain, Myofascial; Neck Muscle Issue; Muscle Tightness; Neckache
Keywords: Dry Needling; Ischemic Compression; Neck Pain
MeSH Terms: conditions — Neck Pain; Myofascial Pain Syndromes | interventions — Dry Needling; Acupressure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling Group (Experimental): Received dry needling through the insertion of fusiform needle for the trigger point release on 3 days a week aimed at pain relief.
  Interventions: Other: Dry Needling
- Ischemic Compression Group (Active Comparator): Received ischemic compression release through thumb pressure for trigger points on 3 days a week.
  Interventions: Other: Dry Needling

INTERVENTIONS:
Other: Dry Needling — Dry Needling includes the insertion of a fine, strong filiform needle without presentation of any pain relieving medicine.
  Ischemic pressure is usually applied to trigger point, in what is known as trigger point therapy, where enough continuous pressure is applied to a trigger point within a tolerable measure of pain, and as discomfort is decreased, extra pressure is gradually applied
  Other Names: Ischemic Compression

SUMMARY:
This randomized control trial was conducted to investigate the efficacy of trigger point dry needling which is a modern treatment intervention compared with ischemic compression release in the patients having neck pain due to myofascial trigger points.

DETAILED DESCRIPTION:
Many treatment protocols have been used in the clinical arena for the improvement of neck pain but un-availability of follow-up studies and lack of evidence of modern treatment interventions are few shortcomings a researcher faces. Thus, a need stands up to address these perspectives for newer treatment strategies. This randomized control trial is conducted to investigate the efficacy of trigger point dry needling which is a modern treatment intervention compared with ischemic compression release in the patients having neck pain due to myofascial trigger points. Findings of this research will assist in creating awareness about better treatment intervention for trigger point release among medical community.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the age group of 20 to 40 years.
* Both Male and female patients.
* Patients presenting with neck pain due to MTrP's.
* The presence of a palpable taut band in the neck region.
* Patients reporting typically referred pain pattern of the MTrP in response to compression.

Exclusion Criteria:

* Patients with any associated comorbidities such as hypertension and diabetes.
* Patients with known history of fibromyalgia syndrome, whiplash injury, cervical spine surgery fracture and cervical radiculopathy.
* Patients with any systemic disease such as rheumatism and tuberculosis or cervical myelopathy and multiple sclerosis.
* Patients with history of myofascial trigger point therapy one month prior to enrollment.
* Patients with non-cooperative attitude, fear or any contraindications to needling.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Change in Pain assessed through Visual Analogue Pain Scale | Data was Collected at Baseline and after week 1,2 & 3.
  To measure the change in terms of betterment or aggravation in the intensity of pain baseline then after week 1,week 2 and after week 3.
Change in degree of disability assessed through Northwick Park Neck Pain Questionnaire. | Data was Collected at Baseline and after week 1,2 & 3.
  To measure change in the intensity of neck pain and the consequent patient disabilities at baseline then after week 1,week 2 and after week 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Bashir Institute of Health Sciences,Bashir General & Dental Hospital, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No